CLINICAL TRIAL: NCT00083798
Title: Family Linkage Study of Obstructive Sleep Apnea (OSA) in Iceland
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1251; 5R01HL072067 (NIH)
Record Dates: First submitted 2004-06-02; First posted 2004-06-04 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Sleep Apnea Syndromes; Lung Diseases; Insulin Resistance
MeSH Terms: conditions — Sleep Apnea Syndromes; Lung Diseases; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples with DNA

SUMMARY:
To study the genetic basis of obstructive sleep apnea using a genealogical approach.

DETAILED DESCRIPTION:
BACKGROUND:

There is family aggregation of obstructive sleep apnea (OSA) as has been shown in the United States, Europe and recently in Iceland. Iceland represents a unique opportunity for genetic research. It is a community that was settled by founders in the 9 th Century, and has developed in relative isolation since that time to its present size of 285,000 persons. Moreover, there is a commitment to record keeping that has allowed deCODE Genetics, who are collaborators on this grant, to develop a computerized genealogy data base that permits the ancestry of individuals to be traced over centuries. This tool, together with the founder nature of the population, makes possible a unique genealogy-driven approach to study the genetics of complex disorders, an approach that has already been successful.

DESIGN NARRATIVE:

The study uses patients with obstructive sleep apnea, who have already been diagnosed in Iceland where large family pedigrees have been identified. The study involves a genome-wide family linkage investigation. This will be conducted with an affected only approach examining allele sharing between affected individuals using 1,100 markers spaced across the genome. The investigators plan to oversample the relatively non-obese subjects providing them the opportunity to evaluate linkage in both relatively non-obese and obese subjects. The linkage study will be complemented with an association study, with unrelated cases and controls, matched for age, gender, and menopausal status. In the association study, they will, as a primary aim, test candidate genes arising from the linkage study and, as a secondary aim, evaluate candidate genes that they believe will be identified in the ongoing Cleveland Family Study. A subset of subjects in both the family linkage and association study will have in-depth phenotyping to determine whether there are sub-phenotypes for this complex disorder and, if so, whether they aggregate in families. This in depth phenotyping will involve upper airway magnetic resonance imaging to evaluate upper airway soft tissue and craniofacial structures, acoustic rhinometry to quantify nasal resistance, a known risk factor for the disorder, and insulin resistance. They will explore whether there are distinct patterns of linkage for the different sub-phenotypes. To accomplish this large genetic study, they have put together the resources of three major organizations--the University of Pennsylvania, the University of Iceland Hospitals, and deCODE Genetics. They propose to leverage the truly unique infrastructure developed by deCODE Genetics, the clinical research programs in sleep apnea at the University of Iceland Hospitals, and the in-depth phenotyping expertise at the University of Pennsylvania to accomplish their goals.

ELIGIBILITY:
Patients with moderate to severe sleep apnea.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sleep apnea patient cohort
Sampling Method: Non-Probability Sample
Enrollment: 2843 (Actual)
Dates: Start 2003-09; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Genotype | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Allan I Pack, M.B., Ch.B., Ph.D., Principal Investigator — University of Pennsylvania